CLINICAL TRIAL: NCT04393935
Title: Advancing Pre-exposure Prophylaxis (PrEP) Access in Pharmacies to Improve PrEP Uptake in Disadvantaged Areas
Brief Title: Pharmacy-based Pre-exposure Prophylaxis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Natalie Crawford, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00106370; 1R34MH119007-01 (NIH)
Record Dates: First submitted 2020-05-15; First posted 2020-05-19 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-04

CONDITIONS: Human Immunodeficiency Virus
Keywords: Behavioral intervention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacy Delivered PrEP Intervention (Experimental): Clients of the study pharmacies who participate in the intervention to receive PrEP through the pharmacy.
  Interventions: Behavioral: Pharmacy Delivered PrEP Intervention

INTERVENTIONS:
Behavioral: Pharmacy Delivered PrEP Intervention — Pharmacy client participants who are eligible and agree to the HIV test will be provided with a pre-packaged kit of a self-administered test for HIV and directed back to the private area of the pharmacy to perform their screening. Pharmacy client participants who test HIV negative will be provided with their results and be given a 30-day prescription for PrEP, culturally appropriate PrEP counseling and a follow-up appointment with a PrEP prescribing physician. Pharmacy client participants will be contacted after 3 months to determine whether they continued PrEP use.

SUMMARY:
The proposed research will develop a culturally appropriate pharmacy pre-exposure prophylaxis (PrEP) delivery model for black men who have sex with men (BMSM) who live in high poverty, racial minority neighborhoods. Increasing access to PrEP through pharmacies has the potential to increase PrEP uptake among BMSM thereby reducing HIV incidence and racial inequities in HIV.

DETAILED DESCRIPTION:
Black men who have sex with men (BMSM) bear the highest burden of HIV in the US. PrEP is the single most effective HIV prevention strategy yet under-utilized among BMSM. When taken every day PrEP can prevent up to 92% of HIV infections. Studies estimate that 48-70% of BMSM are willing to use PrEP, yet, uptake among blacks remains low (~10%). Lower insurance rates among blacks compared to whites may be a barrier to PrEP, but, evidence of insurance rates, as well as prescription payment programs that cover most or all of the costs of PrEP do not completely explain significant disparities in PrEP uptake. Indeed, limited access to PrEP, distrust of physicians and stigma are noted as critical barriers to PrEP that must be improved to reduce HIV.

Neighborhood residence shapes BMSM HIV exposure and access to HIV prevention resources. Census tracts with high HIV had 20% higher poverty and 200% larger MSM populations. High poverty neighborhoods also have the fewest HIV physicians. While most census tracts are within 15 minutes of an HIV physician by car, residents in HIV prevalent areas have low rates of car ownership and commute time more than doubles when traveling by public transportation, which is unavailable in some areas.

There is a strong scientific premise for increasing PrEP delivery in pharmacies for BMSM. About 95% of Americans live within 5 miles of a pharmacy; pharmacies have flexible hours and pharmacists have high credibility with community members. Studies have shown pharmacies can engage with high risk populations including people who inject drugs (PWID) to reduce HIV risk behaviors and provide primary prevention services including immunizations, blood pressure screenings and HIV testing. PrEP has also been sustainably offered in a Seattle pharmacy, but mostly to white MSM (85%). Nevertheless, almost 100% initiated PrEP and 75% followed up for continued PrEP. Following this, Walgreens across the US have offered PrEP through their existing clinics.

Existing pharmacy PrEP models have limited potential for reaching BMSM. In Seattle, state regulations give pharmacists authority to administer biological screenings (HIV, sexually transmitted infections (STIs) and creatinine) and prescribe PrEP. Many states do not have legislation that expand pharmacists' purview in service delivery. Walgreens has overcome this regulatory limitation by using nurse practitioners to screen and prescribe PrEP in their existing clinics. While Collaborative Practice Agreements between pharmacists and physicians are another route to deliver services through pharmacies, they are time-consuming and thus infeasible for community pharmacists in high morbidity neighborhoods who already have a hectic workflow; and for chain pharmacies these partnerships are determined on a corporate rather than individual pharmacy level.

Accomplishing the study aims will be done through three steps: conducting interviews and workflow assessments with stakeholders, developing an intervention to deliver a culturally relevant pharmacy PrEP model, and perform a pilot test to study the delivery model in pharmacies in high poverty, racial minority neighborhoods.

In the pilot test phase, pharmacies will be chosen to test the pharmacy PrEP delivery model by informing pharmacy clients of the study and performing their study activities. Pharmacists and technicians will complete a pharmacy-based HIV prevention training to equip them with the tools needed for optimal PrEP delivery. During the training, pharmacists and technicians will learn how to engage pharmacy clients for recruitment into the study. Black race is not included in the eligibility criteria to avoid profiling and potentially stigmatizing one racial group. However, since the pharmacies selected to be a part of the study are located in racial minority neighborhoods, the researchers anticipate that most customers will be racial minorities. Male sex is also not included in the eligibility criteria. The researchers will be collecting both qualitative and quantitative data to assess the impact of the pharmacy PrEP intervention on the pharmacy environment, personnel, and business flow. Among the pharmacy clients, this study will assess feasibility, acceptability and safety of the intervention activities, satisfaction with the activities and participation in activities without stigmatization, discomfort or harm.

The study pharmacies will deliver the PrEP intervention. Pharmacy client participants will receive a 3-month follow-up phone call to see if they are continuing to use PrEP.

ELIGIBILITY:
Inclusion Criteria:

* Consent to participate in the online screener
* Can speak and read English without any help
* Test negative for HIV
* Agree to receive medication from the pharmacy

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2024-05-11 (Actual); Study Completion 2024-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Crawford, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled through study pharmacies in Atlanta, Georgia, USA. Pharmacy client participant enrollment began May 19, 2022 and all follow-up assessments were completed by May 11, 2024.
Groups:
- Pharmacy Delivered PrEP Intervention: Clients of the study pharmacies who participate in the intervention to receive Pre-exposure Prophylaxis (PrEP) through the pharmacy.
  Pharmacy Delivered PrEP Intervention: Pharmacy client participants who are eligible and agree to the HIV test will be provided with a pre-packaged kit of a self-administered test for HIV and directed back to the private area of the pharmacy to perform their screening. Pharmacy client participants who test HIV negative will be provided with their results and be given a 30-day prescription for PrEP, culturally appropriate PrEP counseling and a follow-up appointment with a PrEP prescribing physician. Pharmacy client participants will be contacted after 3 months to determine whether they continued PrEP use.
Period: Overall Study
Arm/Group | Pharmacy Delivered PrEP Intervention
Started | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pharmacy Delivered PrEP Intervention
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 45
  White | 0
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Continuing PrEP
Description: Participants who were prescribed PrEP through the pharmacy intervention were contacted after 3 months to see if they continued PrEP use.
Time Frame: Month 3
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacy Delivered PrEP Intervention
Number analyzed (Participants) | 49
Participants | 2

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected at the baseline assessment and continued through the final assessment at Month 3, for a total of 3 months.
Description: Information on adverse events was collected only for events related to self-testing or PrEP initiation.
Arm/Group | Pharmacy Delivered PrEP Intervention
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT04393935/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT04393935/ICF_000.pdf